CLINICAL TRIAL: NCT02937155
Title: HSIL/ACIS/Early Cervical Cancer: What Are The Current Causative HPV Subtypes in the Era of HPV Vaccination?
Brief Title: In the Era of the HPV Vaccine, What Are The Current HPV Subtypes Contributing to High Grade Cervical Dysplasia, Adenocarcinoma in Situ, and Early Cervical Cancer?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 53257
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-04

CONDITIONS: HSIL, High-Grade Squamous Intraepithelial Lesions; Adenocarcinoma in Situ; Early Cervical Cancer
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Adenocarcinoma in Situ; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccinated: Patients who have received the HPV vaccine.
- Vaccine Naive: Patients who have not received the HPV vaccine.

SUMMARY:
This study will look at cervical tissue samples in women with abnormal cervical cells to see if the frequency of the HPV 16/18 subtypes has changed in female populations today, after the introduction of the HPV vaccine. It will compare women who have been exposed to the HPV vaccine with those who have not.

DETAILED DESCRIPTION:
The development of cervical dysplasia (precursor to cervical cancer) and cervical cancer requires infection with one of several cancer causing subtypes of the human papilloma virus (HPV). There are over 100 subtypes of HPV, and most are not cancer causing. In the past, North American data has shown that 70% of early cervical cancers were associated with HPV subtypes 16 and/or 18. The first HPV vaccines to be approved protected against the common subtypes of HPV 16 and 18. The traditional HPV vaccination consists of 3-doses administered over a 6 month period.

Since the 8 years after the introduction of the vaccine, there have not been any studies analyzing HPV subtype changes. It is important to determine if the prevalence of the HPV subtypes associated with precancerous and/or early cervical cancer have changed, and what preventative outcomes have arisen from the HPV vaccination. This will have implications regarding the importance and anticipated effects of immunization with the nanovalent vaccine that includes other oncogenic subtypes.

This study will look at tissue samples to see if the frequency of the HPV 16/18 subtypes has changed in female populations today, after the introduction of the HPV vaccine. It will compare women who have been exposed to the HPV vaccine with those who have not.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old
* Presenting with cervical high grade intraepithelial dysplasia (HSIL), adenocarcinoma in situ (ACIS), or early cervical cancer
* Fulfills one of the following two criteria:

Expected to have a cervical biopsy, loop electrosurgical excision procedure (LEEP), or cone biopsy as part of standard of care treatment OR Has already had a cone biopsy of LEEP and the archived tissue is located at Sunnybrook Health Sciences Centre and was taken within two years from the time of consent.

Exclusion Criteria:

* A history of HSIL, ACIS, or early cervical cancer prior to 2010
* Patients who are unable to provide consent
* Women who have had a previous LEEP or cone biopsy and tissue removed is greater than 2 years old, from the time of consent
* women who have had a previous LEEP or cone biopsy and tissue is archived at an outside institution

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women recently diagnosed with either high grade cervical dysplasia, ACIS, on early cervical cancer who present to the Sunnybrook Colposcopy Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-06 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Overall prevalence of HPV subtypes | Baseline
  To determine the prevalence of HPV subtypes in HSIL/ACIS/early cervical cancer in patients who have been exposed or naïve to an HPV vaccine.
Reasons for vaccine failures | Baseline
  A descriptive analysis to explore the potential reasons for HPV vaccine failures in women with HSIL/ACIS/early cervical cancer in patients who have been exposed to an HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Covens, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada